CLINICAL TRIAL: NCT05327270
Title: Pilot, Non-randomized, Open-label Study of Intralesional Nivolumab for High Risk Oral Premalignant Lesions
Brief Title: Non-randomized, Open-label Study of Intralesional Nivolumab for High Risk Oral Premalignant Lesions
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1011; NCI-2022-02940 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab will be given as an injection directly into an oral lesion.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Given by IT
  Other Names: BMS-936558; Opdivo

SUMMARY:
To characterize the safety and tolerability of nivolumab injected intralesionally in patients with high-risk oral premalignant lesions.

DETAILED DESCRIPTION:
OBJECTIVES

Primary objective:

To characterize the safety and tolerability of nivolumab injected intralesionally in patients with high-risk oral premalignant lesions.

Secondary objectives:

To describe the objective response rate (ORR) in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions, according to modified World Health Organization (WHO) criteria.

To describe the pathologic complete response (CR) rate in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions.

To describe the major pathologic response rate in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions.

To evaluate systemic exposure of nivolumab following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions.

To assess the immunogenicity of nivolumab in patients with high-risk oral premalignant lesions.

To establish a recommended dose of intralesional nivolumab for further study in patients with high-risk oral premalignant lesions.

ELIGIBILITY:
Subject Inclusion Criteria:

In order to be eligible for this trial, the subject must:

1. Presence of a treatment naïve, biopsy proven, intraoral premalignant lesion visible from oral cavity.
2. Be willing and able to provide written informed consent for the trial.
3. Be >/= 18 years of age on day of signing informed consent.
4. Be willing to provide tissue, either archive or from a newly obtained oral biopsy.
5. Have a performance status of 0-2 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined in Table 1

   Table 1 Adequate Organ Function Laboratory Values Hematological Absolute neutrophil count (ANC) ≥1,000 /mcL Platelets ≥75,000 / mcL Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
7. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of study therapy through 120 days after the last dose of Nivolumab. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Subject Exclusion Criteria:

The subject must be excluded from the trial if the subject:

1. Is currently participating and receiving study therapy with potential anti-neoplastic activity or has participated in a study of an investigational agent and received study therapy with potential anti-neoplastic activity within 4 weeks of the first dose of treatment.
2. Has a known history of active TB (Bacillus Tuberculosis)
3. Hypersensitivity to nivolumab or any of its excipients.
4. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 2 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 2 or at baseline) from adverse events due to a previously administered agent.
6. Has a known additional malignancy that is progressing or requires active treatment other than adjuvant hormonal therapy. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin or in situ cervical cancer.
7. Has known history of, or any evidence of active, non-infectious pneumonitis.
8. Has an active infection requiring systemic therapy.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of treatment with pembrolizumab, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
12. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the objective response rate (ORR) in index lesions following intralesional injections of nivolumab in patients with high-risk oral premalignant lesions, according to modified World Health Organization (WHO) criteria. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Moran Amit, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT05327270/ICF_000.pdf